CLINICAL TRIAL: NCT00553332
Title: A Phase 2 Study of AZD6244 in Biliary Cancers
Brief Title: Selumetinib in Treating Patients With Biliary Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00251; OSU 07056; OSU-07056; CDR0000573452; N01CM62208 (NIH); N01CM62207 (NIH); NCT01645644 (obsolete NCT alias)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Liver and Intrahepatic Biliary Tract Cancer; Recurrent Extrahepatic Bile Duct Cancer; Unresectable Extrahepatic Bile Duct Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Bile Duct Neoplasms | interventions — AZD 6244

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive oral selumetinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: selumetinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: selumetinib — Given orally
  Other Names: ARRY-142886; AZD6244
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well selumetinib works in treating patients with biliary cancer that cannot be removed by surgery. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (complete response [CR] and partial response [PR]) in patients with unresectable biliary carcinoma treated with AZD6244 (selumetinib).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile of this drug in these patients. II. To evaluate the 6- and 12-month survival, 6-month progression-free survival, and overall survival rates of patients treated with this drug.

III. To correlate genetic mutations, epigenetic silencing, and/or protein levels of RAS/RAF/MEK/ERK signaling pathway activation with therapeutic efficacy of AZD6244 in these patients.

IV. To genotype tumors for the presence of RAS mutations (i.e., NRAS, KRAS, HRAS) and BRAF mutations (e.g., V600E) in biliary tumor samples from these patients.

V. To assess the presence of activation of the MEK1, MEK2, ERK, and/or Akt pathways in tumor samples from these patients.

VI. To assess the epigenetic alterations (i.e., methylation) affecting the level of gene/protein expression of RASSF1A, NORE1A, and NORE1B in tumor samples from these patients.

OUTLINE:

Patients receive oral selumetinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Formalin fixed paraffin-embedded tissue blocks or fresh tissue samples are obtained from all patients prior to treatment. Tissue samples are analyzed by immunohistochemistry for the expression level of target proteins (MEK, p-MEK, ERK, p-ERK, Akt, p-AKT, RASSF1A, NORE1A and NORE1B); PCR for mutational status of target genes RAS, BRAF and EGFR); and in methylation-specific PCR for methylation of target gene promoters (promoters for RASSF1A, NORE1A and NORE1B). Samples are also analyzed by quantitative real-time PCR to compare methylation status. Fresh frozen tissue, when available, is evaluated by Western analysis to measure expression levels of target proteins.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed biliary tract carcinoma

  * Surgically unresectable disease
* Meets any of the following criteria for biliary cancers only:

  * Received ≤ 1 prior systemic anticancer therapy, including chemoembolization
  * Received prior cryotherapy, radiofrequency ablation, ethanol injection, transarterial chemoembolization, or photodynamic therapy AND meets the following criteria:

    * More than 6 weeks have elapsed since any of the prior therapy described above
    * Indicator lesion(s) must be outside the area of prior treatment OR must demonstrate clear evidence of disease progression if the only indicator lesion is inside the prior treatment area
    * Indicator lesion must have clearly distinct edges on CT scan
  * Prior radiotherapy with or without the use of a fluoropyrimidine as a radiosensitizer is allowed, provided more than 12 weeks have elapsed since treatment
* Fresh or paraffin-embedded tissue from tumor blocks must be available for review
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques or > 10 mm by spiral CT scan
* No known brain metastases
* Life expectancy > 12 weeks
* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100%
* ANC ≥ 1,500/μL
* Platelet count ≥ 75,000/μL
* Total bilirubin ≤ 2 times upper limit of normal(ULN)
* AST or ALT ≤ 3 times ULN
* Serum albumin ≥ 2.5 mg/dL
* INR ≤ 1.5 (not receiving anticoagulation therapy)
* Creatinine normal or creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile women must use effective contraception during and for four weeks after the last dose of AZD6244
* Fertile men must use effective contraception during and for 16 weeks after the last dose of AZD6244
* No significant traumatic injury within the past 3 weeks
* No uncontrolled symptoms consistent with encephalopathy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 or its excipient, Captisol®
* No QTc interval > 500 msecs or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., hypokalemia or family history of long QT interval syndrome), including NYHA class III-IV heart failure
* No other malignancy within the past 3 years, except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No refractory nausea and vomiting, chronic gastrointestinal disease (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* No uncontrolled concurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situation that would limit compliance with study requirements
* No malignant hypertension within the past year
* No prior sorafenib or MEK inhibitors
* More than 4 weeks since prior chemotherapy, biologic therapy, or immunotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered to ≤ grade 1 adverse events
* No major surgery within the past 3 weeks
* No other concurrent investigational agents
* No concurrent requirement for medication that can prolong the QT interval
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent consumption of grapefruit or grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, Principal Investigator — Ohio State University
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Michigan Cancer Center (UMCC) Research Base, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Bekaii-Saab T, Phelps MA, Li X, Saji M, Goff L, Kauh JS, O'Neil BH, Balsom S, Balint C, Liersemann R, Vasko VV, Bloomston M, Marsh W, Doyle LA, Ellison G, Grever M, Ringel MD, Villalona-Calero MA. Multi-institutional phase II study of selumetinib in patients with metastatic biliary cancers. J Clin Oncol. 2011 Jun 10;29(17):2357-63. doi: 10.1200/JCO.2010.33.9473. Epub 2011 Apr 25. PMID 21519026

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled to the trial between December 2007 and January 2009
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 29
Completed | 28 (evaluable for response)
Not Completed | 1
Not completed — ineligible, incorrect diagnosis | 1

BASELINE CHARACTERISTICS:
Population: All patients had metastatic disease.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 55.6 [26 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 28
Eastern Cooperative Oncology Group (ECOG) [Number; unit: patients]
  0 (Fully active) | 11
  1 (Restricted activity) | 17
Disease site [Number; unit: patients]
  Intrahepatic | 17
  Gallbladder | 7
  Extrahepatic | 4
Metastasis site [Number; unit: patients]
  Liver only | 7
  Liver and other sites | 16
  Other (soft tissue, lymph nodes and lung) | 5
Number of target lesions [Median (Full Range); unit: lesions] | 4 [1 to 13]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (CR and PR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 8 weeks
Measure: Number; unit: patients
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 25
patients
  Complete Response | 0
  Partial Response | 3

2. Secondary Outcome: Toxicity Profile of AZD6244
Description: Toxicitity will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 3.0
Time Frame: From the time of first treatment with AZD6244, assessed up to 4 weeks
Measure: Number; unit: percent of patients
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 28
percent of patients
  Rash | 90
  Xerostomia | 54
  Nausea | 50

3. Secondary Outcome: Median Progression Free Survival for Patients
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 28
months | 3.7 [3.5 to 4.9]

4. Secondary Outcome: Overall Survival
Time Frame: Up to 12 months
Population: Kaplan-Meier
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 28
months | 9.8 [3.50 to NA] — Too early to reach the upper 95% confidence interval

5. Secondary Outcome: RAS/RAF/MEK/ERK Signaling Pathway Activation
Time Frame: At baseline
Population: Data was not collected and analyzed
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Protein Levels of RAS/RAF/MEK/ERK Signaling Pathway Activation
Description: Measure the proteins levels of RAS/RAF/MEK/ERK signaling pathway activation to AZD6244
Time Frame: At baseline
Population: Only 27 patients had pAKT and pERK performed due to 2 samples not available for analysis
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 28
mg/ml
  pAKT | 1.23 (0.98)
  pERK | 1.36 (1.09)

ADVERSE EVENTS:
Time Frame: All patients were evaluated for toxicity using the NCI Common Toxicity Criteria version 3.0 from the time of their first treatment until the end of treatment.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 28/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=28)
Rash (Skin and subcutaneous tissue disorders) | 25 (25)
Xerostomia (Gastrointestinal disorders) | 15 (15)
Nausea (Gastrointestinal disorders) | 14 (14)
Vomiting (Gastrointestinal disorders) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Bloating (Gastrointestinal disorders) | 12 (12)
Dry Skin (Skin and subcutaneous tissue disorders) | 11 (11)
Dysgeusia (Nervous system disorders) | 8 (8)
Mucositis (Gastrointestinal disorders) | 7 (7)
Flatulence (Gastrointestinal disorders) | 6 (6)
Thrombocytopenia (Injury, poisoning and procedural complications) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less